CLINICAL TRIAL: NCT06127966
Title: The Relationship Between the Preoperative Neutrophil-to-lymphocyte Ratio (NLR) and Postoperative Nausea and Vomiting (PONV) in Lumbar Spine Surgery Patients, as Well as the Impact of Erector Spinae Plane Block on NLR and PONV
Brief Title: The Relationship Between NLR and PONV and ESPB
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Guanghan Wu, Attending physician, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YXLL-KY-2023（101）
Record Dates: First submitted 2023-10-29; First posted 2023-11-13 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Erector Spinae Plane Block; Neutrophil to Lymphocyte Ratio
Keywords: Neutrophil to Lymphocyte Ratio; Postoperative Nausea and Vomiting; erector spinae plane block; Postoperative analgesia; lumbosacral spine surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector Spinae Plane Block group(EA group + EB group) (Experimental): Conventional anesthesia induction, followed by ultrasound-guided erector spinae plane (ESPB) block with 0.5% ropivacaine (20 ml) after anesthesia induction.
  Interventions: Procedure: Erector Spinae Plane Block
- Control group（CA group + CB group) (Sham Comparator): Conventional anesthesia induction, followed by ultrasound-guided injection of 0.9% saline (20 ml) into the erector spinae plane (ESPB) after anesthesia induction.
  Interventions: Procedure: 0.9% physiological saline (20ml) injection under ultrasound-guided Erector Spinae Plane Block (ESPB).

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — The patient assumes a prone position, and the appropriate lumbar vertebral level is identified using ultrasound, based on the preoperative markings of the surgical incision site. After disinfection, the ultrasound probe is placed in the parasagittal direction, 3 centimeters lateral to the midline, to identify the corresponding lumbar transverse process and the overlying erector spinae and latissimus dorsi muscles. Using an in-plane technique, the needle is advanced, and when the needle tip contacts the bony transverse process and there is no blood or gas upon aspiration, 2-3 mL of isotonic saline solution is injected to confirm the correct needle position. Local anesthetic is then injected between the erector spinae muscle and the transverse process. The spread of the local anesthetic in the deep fascial plane within the erector spinae muscle can be visualized using ultrasound.
  Arms: Erector Spinae Plane Block group(EA group + EB group)
Procedure: 0.9% physiological saline (20ml) injection under ultrasound-guided Erector Spinae Plane Block (ESPB). — The patient is placed in a prone position, and the appropriate lumbar vertebral level is determined using ultrasound based on the preoperative markings of the surgical incision site. After disinfection, the ultrasound probe is positioned in the parasagittal direction, 3 centimeters lateral to the midline, to identify the corresponding lumbar transverse process, erector spinae, and latissimus dorsi muscles above it. Using an in-plane technique, the needle is advanced, and when the needle tip contacts the bony transverse process, and there is no blood or gas upon aspiration, 2-3 milliliters of isotonic saline solution are injected to confirm the correct needle position. Subsequently, 20 milliliters of 0.9% physiological saline is injected between the erector spinae muscle and the transverse process. The diffusion of the physiological saline in the deep fascial plane within the erector spinae muscle can be visualized using ultrasound.
  Arms: Control group（CA group + CB group)

SUMMARY:
This study aims to investigate whether preoperative NLR (Neutrophil-to-Lymphocyte Ratio) serves as a biomarker for PONV (Postoperative Nausea and Vomiting). It also examines the impact of erector spinae plane block on NLR and PONV. Furthermore, the research explores the effect of erector spinae plane block on postoperative pain relief in spinal surgery and its influence on the usage of opioid medications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective posterior lumbar spine surgery in a prone position under general anesthesia.
2. ASA classification grades I to II.
3. Age between 18 and 80 years old.
4. Signed the informed consent for this study.

Exclusion Criteria:

1. Preoperative blood transfusion.
2. Uncontrolled systemic diseases.
3. Patients with known uncontrolled systemic inflammatory diseases (e.g., rheumatoid arthritis, lupus, or active infections).
4. Gastrointestinal system disorders.
5. History of antiemetic and anticholinergic drug use.
6. History of adverse reactions related to surgery, deformity correction surgeries, defined as procedures involving instrumentation across three or more levels or aimed at correcting scoliosis or kyphosis.
7. Severe spinal deformities.
8. Infection at the puncture site.
9. Coagulation disorders.
10. Long-term use of sedatives and analgesic drugs before surgery.
11. Patients with mental illness or communication barriers.
12. Allergic to ropivacaine.
13. Participants involved in other clinical studies within the past 3 months.
14. History of previous lumbar surgeries.
15. Subjective unwillingness to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Record nausea and vomiting within the PACU and during the first 24 hours and second 24 hours after surgery. | Within the first 24 hours and the second 24 hours after surgery.
  Patients with a nausea and vomiting score of 1 point or above (0 points = no nausea, 1 point = nausea, 2 points = dry heaving, 3 points = vomiting) are treated with ondansetron as an antiemetic.
Record the need for antiemetic medication within the PACU and during the first 24 hours and the second 24 hours postoperatively. | Within the first 24 hours and the second 24 hours after surgery.
  Record the need for antiemetic medication within the PACU and during the first 24 hours and the second 24 hours postoperatively.
Record the neutrophil count and lymphocyte count on the first day after surgery and calculate the neutrophil-to-lymphocyte ratio (NLR) | Within the first 24 hours.
  The neutrophil count and lymphocyte count and calculate the neutrophil-to-lymphocyte ratio (NLR).

SECONDARY OUTCOMES:
Overall VAS (Visual Analog Scale) pain scores at 2 hours, 6 hours, 12 hours, 24 hours, and 48 hours postoperatively during rest and movement. | At 2 hours, 6 hours, 12 hours, 24 hours, and 48 hours after surgery
  VAS scoring criteria, also known as pain level scoring criteria, use a visual analog method to assess the severity of pain.The VAS (Visual Analog Scale) rating ranges from 0 to 10, with a VAS score of 0 indicating no pain. Scores of 1-3 represent mild pain (pain does not affect sleep), 4-6 indicate moderate pain (pain disrupts sleep), 7-9 correspond to severe pain (unable to fall asleep or waking up due to pain, or unable to sleep), and a score of 10 signifies excruciating pain. The higher the score, the more severe the pain.
Record the time of the patient's initial self-administration of the pain pump during the first 24 hours and the second 24 hours after surgery. | Within the first 24 hours and the second 24 hours after surgery
  Record the time of the patient's initial self-administration of the pain pump during the first 24 hours and the second 24 hours after surgery.
Record the time of the initial press of the patient-controlled analgesia pump. | Within the first 24 hours and the second 24 hours after surgery
  Record the time of the initial press of the patient-controlled analgesia pump.
Record the satisfaction scores for pain management at 24 and 48 hours. | Within the first 24 hours and the second 24 hours after surgery
  Patient satisfaction score refers to the postoperative satisfaction level of the patient, with 0 points indicating dissatisfaction, 1 point indicating fair, 2 points indicating satisfaction, and 3 points indicating very satisfied. The higher the score, the more satisfied the patient is with the treatment outcome.
Record the postoperative awakening time. | Within 24 hours.
  Record the postoperative awakening time.
Record the extubation time after surgery. | Within 24 hours.
  Record the extubation time after surgery.
Postoperative stay in the PACU (Post-Anesthesia Care Unit). | Within 24 hours.
  Postoperative stay in the PACU (Post-Anesthesia Care Unit).
Time of discharge post-surgery. | Within 2 weeks.
  Time of discharge post-surgery.
Document the occurrence rate of opioid-related side effects such as dizziness and urinary retention. | Within 1 week
  Document the occurrence rate of opioid-related side effects such as dizziness and urinary retention.
Measure neutrophil extracellular trap (NETs) formation in serum on the first postoperative day. | At 24 hours after surgery
  Measure neutrophil extracellular trap (NETs) formation in serum on the first postoperative day.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang JJ, Wang Y, Li XF, Chen SS, Wang Y, Sun PY, Yang HK, Shi P, Wu G. The impact of erector spinae plane block on neutrophil-to-lymphocyte ratio and postoperative nausea and vomiting in lumbar spine surgery patients: a protocol for a randomized controlled trial. Front Med (Lausanne). 2025 Aug 28;12:1630821. doi: 10.3389/fmed.2025.1630821. eCollection 2025. PMID 40950965